CLINICAL TRIAL: NCT02553382
Title: Co-administration of Three Complimentary Therapies (Viscous Dietary Fiber, Whole Grain and Ginseng) for Comprehensive Risk Reduction in Type 2 Diabetes Mellitus
Brief Title: Fibre Grain Herb Trial in Type 2 Diabetes
Acronym: FIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-111
Record Dates: First submitted 2015-07-30; First posted 2015-09-17 (Estimated); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Dietary, Herbal (Experimental)
  Interventions: Dietary Supplement: Dietary, Herbal
- Positive Control (Placebo Comparator)
  Interventions: Dietary Supplement: Positive Control

INTERVENTIONS:
Dietary Supplement: Dietary, Herbal — Viscous fibre blend and Salba and American and Korean Red Ginseng capsules
  Arms: Dietary, Herbal
Dietary Supplement: Positive Control — Oat bran blend and wheat bran capsules
  Arms: Positive Control

SUMMARY:
Despite the availability of multiple medications for the treatment of Type 2 diabetes, patients often continue to have difficulty attaining blood glucose targets and managing cardiovascular disease risk factors. Recent trends in non-pharmacological therapy have created a growing public interest in dietary supplements.

Research by this group and others support the benefits of whole grains, viscous dietary fibre and ginseng in the management of diabetes. The current study investigates whether the co-administration of a viscous dietary fibre blend, Salba (a grain rich in omega-3 fatty acids), and 2 varieties of ginseng roots will further improve blood sugar control and cardiovascular disease risk outcomes in individuals with Type 2 diabetes already receiving conventional treatments.

Patients with Type 2 diabetes receiving the recommended intervention in accordance with the Canadian Diabetes Association guidelines will be enrolled in a 6-month clinical study. Half of the participants will be randomly assigned to a 4-component intervention that comprises the co-administration of these four dietary/herbal supplements in addition to their usual treatment regimen; the other half will continue their usual treatment regimen in addition to taking high-oat fiber and wheat bran supplements.

The investigators hypothesize that an intensified, multi-targeted intervention with the addition of these dietary and herb components will further improve long-term blood glucose control and cardiovascular disease risk factors beyond conventional therapy. If this combination of viscous fiber, Salba and ginseng is shown to be beneficial, these remedies could complement current conventional therapy for Type 2 diabetes with the goal to further improve health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes medically diagnosed for at least 6-months prior to randomization
* HbA1c (glycated hemoglobin) between 6.3% and 8.5% at screening
* BMI < 35 kg/m2

Exclusion Criteria:

* Insulin therapy
* Blood pressure ≥ 160/100 mmHg
* Serum triglyceride >4.5mmol/L
* History of major cardiovascular events (stroke or myocardial infarction)
* Gastrointestinal, liver or kidney disease
* Consumption of alcohol >2 drinks/day
* Current tobacco smokers
* Taking the following medications: herbs or supplements that may affect primary or secondary outcomes, monoamine oxidase inhibitors (MAOIs) antidepressants and/or anticoagulant therapy
* Women with hormone sensitive tumors/conditions

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-11; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Baseline to 24 weeks
  Assessed via laboratory analysis

SECONDARY OUTCOMES:
Change in LDL-C | Baseline to 24 weeks
  Assessed via laboratory analysis
Change in 24h ambulatory systolic blood pressure | Baseline to 24 weeks
  Assessed via analysis

OTHER OUTCOMES:
Change in fasting glucose | Baseline to 24 weeks
  Assessed via laboratory analysis
Change in fasting insulin | Baseline to 24 weeks
  Assessed via laboratory analysis
Change in HOMA-IR | Baseline to 24 weeks
  Assessed via laboratory analysis
Change in total cholesterol | Baseline to 24 weeks
  Assessed via laboratory analysis
Change in triglycerides | Baseline to 24 weeks
  Assessed via laboratory analysis
Change in HDL-C | Baseline to 24 weeks
  Assessed via laboratory analysis
Change in total cholesterol:HDL-C | Baseline to 24 weeks
  Assessed via laboratory analysis
Change in Non-HDL-C | Baseline to 24 weeks
  Assessed via laboratory analysis
Change in Apo-B | Baseline to 24 weeks
  Assessed via laboratory analysis
Change in 24h diastolic BP | Baseline to 24 weeks
  Assessed via analysis
Change in office systolic BP | Baseline to 24 weeks
  Assessed via analysis
Change in office diastolic BP | Baseline to 24 weeks
  Assessed via analysis
Change in central systolic BP | Baseline to 24 weeks
  Assessed via analysis
Change in central diastolic BP | Baseline to 24 weeks
  Assessed via analysis
Change in Augmentation index at heart rate 75 bpm | Baseline to 24 weeks
  Assessed via analysis
Change in Hs-CRP | Baseline to 24 weeks
  Assessed via laboratory analysis

CONTACTS AND LOCATIONS:
Locations (2):
- St. Michael's Hopsital, Toronto, Ontario, Canada
- Clinical Centre Vuk Vrhovac, Merkur Hospital, Zagreb, Croatia

REFERENCES:
- [Derived] Zurbau A, Smircic Duvnjak L, Magas S, Jovanovski E, Miocic J, Jenkins AL, Jenkins DJA, Josse RG, Leiter LA, Sievenpiper JL, Vuksan V. Co-administration of viscous fiber, Salba-chia and ginseng on glycemic management in type 2 diabetes: a double-blind randomized controlled trial. Eur J Nutr. 2021 Sep;60(6):3071-3083. doi: 10.1007/s00394-020-02434-7. Epub 2021 Jan 24. PMID 33486572